CLINICAL TRIAL: NCT05472597
Title: Continuation of the nuMoM2b Heart Health Study
Acronym: nuMoM2b-HHS2
Status: Enrolling by invitation | Type: Observational
Sponsor: RTI International (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Northwestern University (Other); Ohio State University (Other); Cedars-Sinai Medical Center (Other); Case Western Reserve University (Other); Columbia University (Other); ChristianaCare (Other); Indiana University (Other); University of Pittsburgh (Other); University of California, Irvine (Other); University of Utah (Other); University of Pennsylvania (Other); Intermountain Health Care, Inc. (Other); University of Michigan (Other); West Virginia University (Other); Old Dominion University (Other)
Responsible Party: Principal Investigator, Becky McNeil, Senior Research Statistician, RTI International
Other Study IDs: 00047665; U01HL145358 (NIH)
Record Dates: First submitted 2022-07-07; First posted 2022-07-25 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; Adverse Pregnancy Outcomes; Stillbirth; Small for Gestational Age; Preterm Birth; Hypertensive Diseases of Pregnancy; Gestational Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Stillbirth; Premature Birth; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We are collecting whole blood, serum, plasma, buffy coat, and urine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- nuMoM2b Heart Health Study Cohort: A large and diverse (both geographically and demographically) group of adult women enrolled and richly phenotyped during their first pregnancy, with data and biospecimens prospective collected thereafter.

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of mortality and morbidity in U.S. women at all ages, and large knowledge gaps exist in CVD predictive and preventative strategies for women. The nuMoM2b Heart Health Study (nuMoM2b-HHS) has followed a demographically diverse cohort of women enrolled and richly phenotyped during their first pregnancy, with data and biospecimens prospectively collected for up to 7 years thereafter. The overarching scientific goal of this study is to define the relationship between adverse pregnancy outcomes (APOs) and CVD to optimize CVD prediction, prevention, and treatment strategies for women. Continued follow-up of this observational cohort, building on a foundation of existing high-quality data, biospecimens, and administrative structures with a robust framework for ancillary study development and implementation, provides a unique opportunity to address knowledge gaps regarding the early mechanisms and trajectory of CVD in women.

DETAILED DESCRIPTION:
The Continuation of nuMoM2b Heart Health Study (nuMoM2b-HHS2) will include prospectively collected longitudinal data on CVD risk factors and early clinical manifestations of CVD, the study's primary outcomes of interest. Measures completed during semiannual follow-ups will include 1) self-reported interval medical history, including medications and substance use; 2) interval pregnancy and postpartum history; 3) interval CVD events, conditions, and diagnostic and therapeutic procedures including CVD death, myocardial infarction (MI), stroke, transient ischemic attack (TIA), pulmonary embolism (PE), deep vein thrombosis (DVT), peripheral vascular disease, kidney disease, hypertension, diabetes, hyperlipidemia, and associated hospitalizations and procedures.

During a study visit in years 3-6, the participant's blood pressure, pulse rate, weight, height, and body measurements will be recorded. During the visit, a fasting blood draw and clean-catch urine specimen will be collected. Aliquots of whole blood, plasma, serum, and urine will be stored at the biorepository; these will be analyzed for CVD measures of lipids, triglycerides, and glucose, among others. Measures of behavioral risk factors, including nutrition, physical activity, and stress will also be completed.

Ancillary studies will expand data collection during the follow-up contacts and in-person visit, and add to the planned contact schedule, to permit the effective targeting of knowledge gaps required to optimize predictive and preventative strategies. Some ancillary studies will only rely on extant data, while others will require de novo data collection during the planned follow-up contacts and/or in-person visits (or participation in additional in-person visits).

ELIGIBILITY:
Inclusion Criteria for nuMoM2b-HHS2 interval contact (telephone interview or web-based self-administered survey):

* Completed one or more interval contacts during the nuMoM2b Heart Health Study.
* Able to speak or read in English or Spanish.

Exclusion Criteria for nuMoM2b-HHS2 interval contact (telephone interview or web-based self-administered survey):

* Withdrawal from study.

Inclusion Criteria for nuMoM2b-HHS2 study visit:

* Completed one or more interval contacts during the nuMoM2b Heart Health Study.
* At least 18 years of age.
* Self-report of at least 3 months postpartum from any subsequent pregnancy.
* Provision of signed informed consent for the HHS2 study visit.
* Able to speak or read English or Spanish.

Exclusion Criteria for nuMoM2b-HHS2 study visit:

* Current pregnancy.
* Withdrawal from study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All nuMoM2b-HHS2 cohort participants will be female. Males were excluded from the original nuMoM2b study because the focus of the study was on the relationship between pregnancy and CVD risk and events.
Study Population: The original nuMoM2b cohort consisted of an ethnically and racially diverse group of pregnant women aged 13 or over who had not had a pregnancy lasting 20 weeks or more, enrolled during the first trimester. Overall, 62% of the nuMoM2b-HHS participants are non-Hispanic white, 14% non-Hispanic black, 16% Hispanic, and 8% mixed race or other. The socio-demographics on the nuMoM2b-HHS participants vary substantially by clinical site, contributing to a rich degree of diversity within the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 4048 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypertension (130/80 mmHg) | Assessed during the HHS2 in-person visit, 8-16 years after the index pregnancy.
  Measured blood pressure > 130/80 mmHg, use of antihypertensive medication, or self-report of a hypertension clinical diagnosis
Incidence of diabetes | Assessed during the HHS2 in-person visit, 8-16 years after the index pregnancy.
  Measured hemoglobin A1c GE 6.5%, fasting blood glucose GE 126 mg/dL, use of blood sugar lowering medication, or self-report of a diabetes clinical diagnosis
Incidence of obesity | Assessed during the HHS2 in-person visit, 8-16 years after the index pregnancy.
  Measured BMI GE 30 kg/m^2
Incidence of metabolic syndrome | Assessed during the HHS2 in-person visit, 8-16 years after the index pregnancy.
  Per the American Heart Association standard definition: Any three of the following five - 1) waist circumference > 35 inches (88 cm) for non-Asians and > 31.5 inches (80 cm) for Asians; 2) triglycerides > 150 mg/dL or medication treatment for high triglycerides; 3) high density lipoprotein (HDL) < 50 mg/dL or medication treatment for low HDL; 4) a serum glucose ≥ 100 mg/dL or a diagnosis of diabetes mellitus; 5) systolic blood pressure (SBP) ≥ 130 mmHg or diastolic blood pressure (DBP) ≥ 85 mmHg, or medication treatment for hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: George Saade, MD, Principal Investigator — Old Dominion University; Phillip Greenland, MD, Principal Investigator — Northwestern University; Rebecca McNeil, PhD, Principal Investigator — RTI International
Locations (14):
- United States (14):
  - University of California, Irvine Medical Center, Orange, California
  - Christiana Care Health Services, Newark, Delaware
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Columbia University Medical Center, New York, New York
  - The MetroHealth System, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - UPMC Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Hospital, Provo, Utah
  - University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available through an NIH data repository.